CLINICAL TRIAL: NCT03185650
Title: Evaluation of Regional Lung Deposition of Inhaled Saline Using the Trans-Nasal Pulmonary Aerosol Delivery Device in Healthy, Non-Smoking Adult Subjects
Brief Title: Evaluation of Regional Lung Deposition of Inhaled Saline Using the tPAD Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Parion Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16-2124
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-07

CONDITIONS: Lung Diseases
Keywords: Healthy Volunteers
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: Healthy subjects will use each nebulizer device in random order at separate study visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- tPAD, then PARI LC Star Nebulizer (Other): tPAD device delivering 14% HS labelled with technetium-99m sulfur colloid particles separated by 2-28 days and then PARI LC delivering 7% HS labeled with technetium-99m sulfur colloid particles.
  Interventions: Device: tPAD Device; Device: PARI LC Star Nebulizer
- PARI LC Star Nebulizer, then tPAD (Other): PARI LC delivering 7% HS labelled with technetium-99m sulfur colloid particles separated by 2-28 days and then tPAD device delivering 14% HS labelled with technetium-99m sulfur colloid particles
  Interventions: Device: tPAD Device; Device: PARI LC Star Nebulizer

INTERVENTIONS:
Device: tPAD Device — A novel, transnasal aerosol generator
Device: PARI LC Star Nebulizer — Standard oral nebulizer

SUMMARY:
Purpose: Characterize the depositional attributes of a specialized trans-nasal aerosol delivery device in healthy people using clinical measurements of mucociliary clearance.

Procedures (methods): 14% hypertonic saline (HS) aerosol containing the radio tracer Tc99m-sulfur colloid will be delivered via the tPAD and compared to the well characterized PARI LC Star nebulizer (7% HS) using planar gamma scintigraphy (i.e. particle clearance). The fraction of sulfur colloid particles that clear over the ensuing 24 hours with each device will indicate the fraction deposited in conducting airways.

DETAILED DESCRIPTION:
Purpose: This is an early device characterization study to define the fraction of delivered aerosol generated by a novel nebulizer (tPAD) that deposits in conducting airways.

Design: Open label, cross-over design, using a standard oral nebulizer (PARI LC Star) as a comparator. The order of visits will be randomized.

Methods: Gamma scintigraphy will be performed following use of each device on separate study visits.

Primary Outcome: Fraction of inhaled particles that clears over 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 to 65 years (inclusive), and with a body mass index (BMI) < 30 kg/m2.
2. Non-pregnant female subjects must be either not sexually active, post-menopausal, surgically sterilized, or agree to use an appropriate "double-barrier" method (such as a diaphragm and condom); or, must currently be using a prescribed transdermal, injection, implant, or oral contraceptive during study participation.
3. Subjects who are in good health, as determined by a medical history and examination.
4. Subjects who have normal lung function with a FEV1 ≥80% predicted and a FEV1/FVC >70%.
5. Subjects who are capable of providing written informed consent in English to participate in the study.

Exclusion Criteria:

1. Subjects who have evidence of an upper or lower respiratory infection or clinically significant illness at entry or within 14 days of the start of dosing.
2. Subjects with lung diseases as defined by a FEV1 <80% or a FEV1/FVC <70%
3. Subjects on inhaled medications, such as short or long acting bronchodilators or inhaled corticosteroids, will be excluded.
4. Subjects with a history of allergy or intolerance to albuterol or hypertonic saline.
5. Subjects with active chronic or acute rhinosinusitis or other nasal or sinus abnormality or disease.
6. Subjects who have a present history of any clinically significant neurologic, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological disorder or disease, substance abuse, or any other major disorder or disease.
7. Subjects who have had radiation exposure within the past year that would cause them to exceed Federal Regulations of 15 Rem annually by participating in this study. The study team will determine this.
8. Subjects with a history of smoking within the last 3 months.
9. Subjects with a positive pregnancy test or who are pregnant or are nursing.
10. Subjects who, in the opinion of the Principal Investigator, should not participate in the study.
11. Subjects with a BMI >30 kg/m2
12. Subjects who are taller than Height >6'2"
13. Subjects who have facial hair that they are not willing to shave

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
24-hour clearance fraction | 24 hours
  The percentage of initially deposited aerosol particles that clear over 24 hours will be measured with gamma scintigraphy after 24 hours

SECONDARY OUTCOMES:
Central:Peripheral Deposition Ratio | 0-4 minutes after deposition
  The ratio of labelled particles initially deposited in the central and peripheral lung zones will be assessed to characterize aerosol targeting of the lung

CONTACTS AND LOCATIONS:
Overall Officials: Scott Donaldson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No